CLINICAL TRIAL: NCT06206135
Title: Multicenter, Open, Prospective, 48 Weeks, Observational Study in the Real-world to Evaluate the Safety and Efficacy of Nephoxil Capsule for Treatment of Hyperphosphatemia in Chronic Kidney Disease Patients on Dialysis
Brief Title: Multicenter, Open, Prospective, 48 Weeks, Observational Study ,Evaluate the Safety and Efficacy of Nephoxil Capsule
Status: Recruiting | Type: Observational
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Other Study IDs: KKKR-Nephoxil OS-01
Record Dates: First submitted 2023-12-17; First posted 2024-01-16 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Population Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 48 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- low-dose group: initial dose 1.5 g/day
  Interventions: Drug: the low-dose group (1.5 g/day) or the standard-dose group (4 g/day)
- standard-dose group: initial dose 4 g/day
  Interventions: Drug: the low-dose group (1.5 g/day) or the standard-dose group (4 g/day)

INTERVENTIONS:
Drug: the low-dose group (1.5 g/day) or the standard-dose group (4 g/day) — The initial dose of Nephoxil capsules for the subjects participating in this study shall be determined at the investigator's discretion, and subjects shall be classified into either the low-dose group (1.5 g/day) or the standard-dose group (4 g/day) according to the initial dose. It will be conducted with 13 visits over 48 weeks.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Nephoxil capsule administration for the improvement of hyperphosphatemia in CKD patients undergoing hemodialysis under actual conditions of routine medical care.

DETAILED DESCRIPTION:
This study is a prospective observational study, and only observable information is collected during Visits 1 to 13 of the subjects' routine outpatient visits. Therefore, no further visits related to this study are planned, and all treatments, examinations, and evaluations necessary for the subjects shall be conducted at the discretion of the investigator.

The initial dose of Nephoxil capsules for the subjects participating in this study shall be determined at the investigator's discretion, and subjects shall be classified into either the low-dose group (1.5 g/day) or the standard-dose group (4 g/day) according to the initial dose. During the observation period, dose titration within 1 g may be performed at the investigator's discretion, and in such cases, the maximum dose per day shall not exceed 6 g.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 19 years of age or older as of the ICF date
2. CKD patients undergoing hemodialysis to whom Nephoxil capsule shall be administered for the first time for the treatment of hyperphosphatemia as per the determination of the investigator
3. Patients who voluntarily decide to participate in this study and complete the ICF

Exclusion Criteria:

1. Those who fall under the "Do not administer to the following patients" criteria according to Nephoxil capsule indication approval
2. Those who require concomitant administration of aluminum-containing medication
3. Others determined by the investigator to be unsuitable for participation in this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hyperphosphatemia in patients with CKD undergoing hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ratio of reached target serum phosphorus level (3.5 - 5.5 mg/dL) at week 48 | 48 weeks
  Ratio of reached target serum phosphorus level (3.5 - 5.5 mg/dL) at week 48

SECONDARY OUTCOMES:
Ratio of subjects whose average serum phosphorus levels at Weeks 40, 44, and 48 reached the target serum phosphorus level (3.5 - 5.5 mg/dL) | 40 ~ 48 weeks
  Ratio of subjects whose average serum phosphorus levels at Weeks 40, 44, and 48 reached the target serum phosphorus level (3.5 - 5.5 mg/dL)
Mean change from baseline to week 48 in serum phosphorus level | 48 weeks
  Mean change from baseline to week 48 in serum phosphorus level
Initial dose retention period | Up to 48weeks
  Initial dose retention period

CONTACTS AND LOCATIONS:
Overall Officials: hyeokjun choi, Study Director — Kyowa Kirin Korea Co., Ltd.
Locations (1):
- Jesus Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided